CLINICAL TRIAL: NCT02441946
Title: neoMONARCH: A Phase 2 Neoadjuvant Trial Comparing the Biological Effects of 2 Weeks of Abemaciclib (LY2835219) in Combination With Anastrozole to Those of Abemaciclib Monotherapy and Anastrozole Monotherapy and Evaluating the Clinical Activity and Safety of a Subsequent 14 Weeks of Therapy With Abemaciclib in Combination With Anastrozole in Postmenopausal Women With Hormone Receptor Positive, HER2 Negative Breast Cancer
Brief Title: A Neoadjuvant Study of Abemaciclib (LY2835219) in Postmenopausal Women With Hormone Receptor Positive, HER2 Negative Breast Cancer
Acronym: neoMONARCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15805; I3Y-MC-JPBY (Other: Eli Lilly and Company); 2014-005486-75 (EudraCT Number)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2015-05-08; First posted 2015-05-12 (Estimated); Results first posted 2018-01-30 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer; Hormone Receptor Positive Tumor; Early-Stage Breast Carcinoma
Keywords: cyclin-dependent kinase (CDK) 4/6 inhibitor; CDK 4 and 6 inhibitor
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib; Loperamide; Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Abemaciclib + Anastrozole (Experimental): Abemaciclib (150 milligrams [mg]) was given orally every 12 hours (Q12H) plus anastrozole (1 mg) orally once daily (QD) for 2 weeks. Loperamide was given as a prophylaxis for 4 weeks and then at physician discretion.
  All participants received abemaciclib (150 mg) orally Q12H plus anastrozole (1 mg) QD for an additional 14 weeks. Total treatment duration was 16 weeks.
  Interventions: Drug: Abemaciclib; Drug: Loperamide; Drug: Anastrozole
- Abemaciclib (Experimental): Abemaciclib (150 mg) was given orally Q12H for 2 weeks. Loperamide was given as a prophylaxis for 4 weeks and then at physician discretion.
  All participants received abemaciclib (150 mg) orally Q12H plus anastrozole (1 mg) QD for an additional 14 weeks. Total treatment duration was 16 weeks.
  Interventions: Drug: Abemaciclib; Drug: Loperamide; Drug: Anastrozole
- Anastrozole (Active Comparator): Anastrozole (1 mg) is given orally QD for 2 weeks.
  All participants received abemaciclib (150 mg) orally Q12H plus anastrozole (1 mg) QD for an additional 14 weeks. Loperamide was given as a prophylaxis for the first 2 weeks of the combination treatment and then at physician discretion. Total treatment duration was 16 weeks.
  Interventions: Drug: Abemaciclib; Drug: Loperamide; Drug: Anastrozole

INTERVENTIONS:
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219
Drug: Loperamide — Administered orally
Drug: Anastrozole — Administered orally

SUMMARY:
The purpose of this study is to evaluate the biological effects of abemaciclib in combination with anastrozole and compare those to the effects of abemaciclib alone and anastrozole alone in the tumors of postmenopausal women with hormone receptor positive (HR+), human epidermal growth factor receptor 2 (HER2) negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have postmenopausal status.
* Adenocarcinoma of the breast.
* Breast tumor ≥1 centimeter (cm) in diameter, HR+, HER2-.
* Neoadjuvant endocrine monotherapy is deemed to be a suitable therapy.
* Primary breast cancer that is suitable for baseline core biopsy.
* Have adequate organ function.

Exclusion Criteria:

* Bilateral invasive breast cancer.
* Metastatic breast cancer (local spread to axillary lymph nodes is permitted).
* Inflammatory breast cancer.
* Prior systemic therapy or radiotherapy for invasive or non-invasive breast cancer in the same breast as currently being treated.
* Prior radiotherapy to the ipsilateral chest wall for any malignancy.
* Prior anti-estrogen therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08-16 (Actual); Study Completion 2018-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (66):
- United States (27):
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - University of California-San Diego, La Jolla, California
  - SMO TRIO -Translational Research, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Cancer Care Associates Medical Group, Redondo Beach, California
  - Sansum Medical Research Foundation, Santa Barbara, California
  - Central Coast Medical Oncology Corporation, Santa Monica, California
  - Stanford University, Stanford, California
  - SMO Pharmatech Oncology Inc, Denver, Colorado
  - St Mary's Hospital Regional Cancer Center, Grand Junction, Colorado
  - Holy Cross Hospital Inc., Fort Lauderdale, Florida
  - Memorial Regional Hospital/Joe Dimaggio Childrens Hospital, Hollywood, Florida
  - Oncology and Radiation Associates, Miami, Florida
  - Orlando Health, Inc, Orlando, Florida
  - Florida Cancer Research Institute, Plantation, Florida
  - Northeast Georgia Cancer Care, LLC, Athens, Georgia
  - Georgia Regents University, Augusta, Georgia
  - Kaiser Foundation Hospitals, Honolulu, Hawaii
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - Nebraska Hematology-Oncology, Lincoln, Nebraska
  - Weill Cornell Medical College, New York, New York
  - St. Charles Health System, Bend, Oregon
  - The West Clinic, Germantown, Tennessee
  - Millennium Oncology, Houston, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Columbia Basin Hematology & Oncology, Kennewick, Washington
- Austria (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Graz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Innsbruck
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Vienna
- Belgium (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Edegem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Hasselt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Namur
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Yvoir
- Canada (2):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Montreal
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Ottawa
- Germany (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Erlangen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Essen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Esslingen am Neckar
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Freiburg im Breisgau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Fürth
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Ludwigsburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Tübingen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Ulm
- Italy (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Napoli
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Padua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Piacenza
- Netherlands (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Maastricht
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Rotterdam
- South Korea (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Daegu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Gangnam-gu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Seodaemun-gu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seongbuk-gu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seongnam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Songpa-gu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Ulsan
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Badajoz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Lleida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Málaga
- Taiwan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Changhua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Taipei

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Franzoi MA, Lambertini M, Ceppi M, Bruzzone M, de Azambuja E. Implication of body mass index (BMI) on the biological and clinical effects of endocrine therapy plus abemaciclib as neoadjuvant therapy for early breast cancer patients. Breast Cancer Res Treat. 2022 Apr;192(2):457-462. doi: 10.1007/s10549-022-06525-3. Epub 2022 Jan 25. PMID 35076812
- [Derived] Hurvitz SA, Martin M, Press MF, Chan D, Fernandez-Abad M, Petru E, Rostorfer R, Guarneri V, Huang CS, Barriga S, Wijayawardana S, Brahmachary M, Ebert PJ, Hossain A, Liu J, Abel A, Aggarwal A, Jansen VM, Slamon DJ. Potent Cell-Cycle Inhibition and Upregulation of Immune Response with Abemaciclib and Anastrozole in neoMONARCH, Phase II Neoadjuvant Study in HR+/HER2- Breast Cancer. Clin Cancer Res. 2020 Feb 1;26(3):566-580. doi: 10.1158/1078-0432.CCR-19-1425. Epub 2019 Oct 15. PMID 31615937
- See also: Click here for more information about this study: A Neoadjuvant Study of Abemaciclib (LY2835219) in Postmenopausal Women With Hormone Receptor Positive, HER2 Negative Breast Cancer — http://www.lillytrialguide.com/EN-us/studies/cancer/jpby

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who had progressive disease at the end of the study but off study drug were considered to have completed the study. Participants were randomized to anastrozole, or abemaciclib, and abemaciclib + anastrozole in cycle 1. All participants received abemaciclib + anastrozole post cycle 1.
Groups:
- Abemaciclib + Anastrozole: Participants were given 150 milligram (mg) of abemaciclib orally every 12 hours (Q12H) plus 1 mg of anastrozole orally once daily (QD) for 2 weeks.
  All participants received 150 mg of abemaciclib orally Q12H plus 1 mg of anastrozole orally QD for an additional 14 weeks.
  Total treatment duration was 16 weeks.
- Abemaciclib: Participants received 150 mg of abemaciclib orally Q12H for 2 weeks.
  All participants received 150 mg of abemaciclib orally Q12H plus 1 mg of anastrozole QD for an additional 14 weeks.
  Total treatment duration was 16 weeks.
- Anastrozole: Participants received 1 mg of anastrozole orally QD for 2 weeks.
  All participants received 150 mg of abemaciclib orally Q12H plus 1 mg of anastrozole orally QD for an additional 14 weeks.
  Total treatment duration was 16 weeks.
Period: Cycle 1 Period 1 (2 Weeks)
Arm/Group | Abemaciclib + Anastrozole | Abemaciclib | Anastrozole
Started | 74 | 76 | 74
Received at Least One Dose of Study Drug | 74 | 75 (1 participant did not receive drug due to an error in randomization.) | 74
Completed | 72 | 71 | 74
Not Completed | 2 | 5 | 0
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0
Not completed — Never Treated | 0 | 1 | 0
Period: Cycle 2-5 Period 2 (14 Weeks)
Arm/Group | Abemaciclib + Anastrozole | Abemaciclib | Anastrozole
Started | 217 (All 217 participants were assigned to abemaciclib + anastrozole post cycle 1.) | 0 (All 217 participants were assigned abemaciclib + anastrozole post cycle 1.) | 0 (All 217 participants were assigned abemaciclib + anastrozole post cycle 1.)
Received at Least One Dose of Study Drug | 217 | 0 | 0
Progressive Disease | 5 | 0 | 0
Completed | 190 | 0 | 0
Not Completed | 27 | 0 | 0
Not completed — Adverse Event | 15 | 0 | 0
Not completed — Noncompliance with study drug | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Protocol Deviation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 0 | 0
Period: Extension Period (8 Weeks)
Arm/Group | Abemaciclib + Anastrozole | Abemaciclib | Anastrozole
Started | 42 (All participants who did not discontinue continued to the extension period.) | 0 | 0
Completed | 40 | 0 | 0
Not Completed | 2 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Abemaciclib + Anastrozole: Participants were given 150 mg of abemaciclib orally Q12H plus 1 mg of anastrozole orally QD for 2 weeks.
  All participants received 150 mg of abemaciclib orally Q12H plus 1 mg of anastrozole orally QD for an additional 14 weeks.
  Total treatment duration was 16 weeks.
- Total: Total of all reporting groups
Arm/Group | Abemaciclib + Anastrozole | Abemaciclib | Anastrozole | Total
Number analyzed (Participants) | 74 | 76 | 74 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (8.4) | 63.8 (7.9) | 64.9 (8.4) | 64.2 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 76 | 74 | 224
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 5 | 19
  Not Hispanic or Latino | 61 | 61 | 60 | 182
  Unknown or Not Reported | 7 | 7 | 9 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 12 | 16 | 16 | 44
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 5 | 1 | 2 | 8
  White | 55 | 57 | 55 | 167
  More than one race | 1 | 1 | 1 | 3
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 0 | 3 | 1 | 4
  Austria | 10 | 4 | 12 | 26
  Netherlands | 1 | 0 | 2 | 3
  Belgium | 5 | 2 | 4 | 11
  United States | 26 | 28 | 26 | 80
  Taiwan | 5 | 7 | 11 | 23
  South Korea | 5 | 7 | 2 | 14
  Italy | 4 | 3 | 4 | 11
  Germany | 5 | 6 | 4 | 15
  Spain | 13 | 16 | 8 | 37
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants]
  0 (Fully Active) | 69 | 70 | 63 | 202
  1 (Restricted, able to do light sedentary work) | 5 | 5 | 10 | 20
  Unreported | 0 | 1 | 1 | 2
Ki67 at Baseline [Mean (Standard Deviation); unit: Percent Cells Positive] — Tumor tissue collected through a core biopsy at baseline and at the end of cycle 1 was used to determine Ki67 expression. Ki67 expression is defined as the percent of cells staining positive by validated central assay.
  Percent Cells Positive | 27.24 (13.56) | 27.88 (12.13) | 26.86 (12.32) | 27.33 (12.63)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to 2 Weeks in Ki67 Expression
Description: Tumor tissue collected through a core biopsy at baseline and at the end of cycle 1 was used to determine Ki67 expression. Ki67 expression is defined as the percent of cells staining positive by validated central assay.
Time Frame: Baseline, 2 Weeks
Population: All randomized participants who received at least one dose of study drug and a valid baseline Ki67 measurement of at least 5% and a valid 2-week measurement of any magnitude.
Measure: Geometric Mean (90% Confidence Interval); unit: Percent Change
Arm/Group | Abemaciclib + Anastrozole | Abemaciclib | Anastrozole
Number analyzed (Participants) | 59 | 52 | 56
Percent Change | -92.86 [-94.82 to -90.16] | -90.52 [-93.12 to -86.93] | -62.78 [-72.99 to -48.71]
Statistical Analysis 1: Comparison: Abemaciclib + Anastrozole vs Anastrozole; Test type: Superiority; p < 0.001, t-test, 1 sided; Ratio of Geometric Means = 0.19, 90% CI 2-sided [0.13 to 0.28]
Statistical Analysis 2: Comparison: Abemaciclib vs Anastrozole; Test type: Superiority; p < 0.001, t-test, 1 sided; Ratio of Geometric Means = 0.25, 90% CI 2-sided [0.17 to 0.38]

2. Secondary Outcome: Percentage of Participants With Pathologic Complete Response (pCR)
Description: pCR is defined as absence of invasive cancer in the breast and sampled regional lymph nodes.
Time Frame: From Start of Treatment Up to 16 Weeks
Population: All participants who received combination treatment post cycle 1 and had evaluable pCR data. Radiological/surgery assessments occurred at the start of treatment and at the end of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Abemaciclib + Anastrozole
Number analyzed (Participants) | 190
percentage of participants | 3.7

3. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR): Clinical Objective Response
Description: Clinical objective response is defined as the percentage of participants with the best overall response rate (ORR) with a best OR of CR or PR, according to Response Evaluation Criteria in Solid Tumors Criteria (RECIST) v1.1. ORR is recorded from the start of the study treatment until the earliest of objective progression or start of new anticancer therapy. A responder depends on target and non-target disease and the appearance of new lesions. CR is defined as the disappearance of all non-target lesions. PR is at least a 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters. All lymph nodes are non-pathological or normal in size (<10mm short axis). Progressive disease (PD) is a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study, a relative increase of 20%, the sum must also demonstrate an absolute increase of 5 mm.
Time Frame: From Start of Treatment to Objective Progression or Start of New Anticancer Therapy (Up to 16 Weeks)
Population: All participants who received combination treatment post cycle 1. Radiological/surgery assessments occurred at the start of treatment and at the end of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Abemaciclib + Anastrozole
Number analyzed (Participants) | 224
percentage of participants | 53.6

4. Secondary Outcome: Percentage of Participants With Complete Radiologic Response or Partial Radiological Response: Radiological Response
Description: Radiological response is the percentage of participants with CR or, PR according to RECIST v.1.1. A responder is defined as any participant who exhibits a CR or PR. CR is the disappearance of all target lesions. PR is a 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters. PD is 20% increase in the sum of diameters of target lesions taking as reference the smallest sum and the appearance of 1 or more new lesions.
Time Frame: From Start of Treatment to Objective Progression or Start of New Anticancer Therapy (Up to 16 Weeks)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Abemaciclib + Anastrozole
Number analyzed (Participants) | 224
percentage of participants | 46.4

5. Secondary Outcome: Change From Baseline to Week 2 in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30)
Description: EORTC QLQ-C30 v3.0 was a self-administered questionnaire with multidimensional scales that measures 5 functional domains (physical, role, emotional, cognitive, or social functioning), global health status and symptom scales of fatigue, pain, nausea/vomiting, dyspnea, insomnia, appetite loss, constipation, diarrhea, or financial difficulties. A linear transformation is applied to standardize the raw scores to range between 0 and 100 per developer guidelines. For functional domains and global health status, higher scores represent a better level of functioning. For symptoms scales, higher scores represented a greater degree of symptoms.
Time Frame: Baseline, 2 Weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable data for EORTC QLQ.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Abemaciclib + Anastrozole | Abemaciclib | Anastrozole
Number analyzed (Participants) | 74 | 76 | 74
units on a scale
  Global Health Status: number analyzed (Participants) | 62 | 66 | 69
  Global Health Status | -9.5 (17.9) | -7.6 (18.1) | -2.3 (13.4)
  Physical Functioning: number analyzed (Participants) | 62 | 66 | 69
  Physical Functioning | -3.2 (10.2) | -5.5 (12.6) | -0.3 (7.5)
  Role Functioning: number analyzed (Participants) | 62 | 66 | 69
  Role Functioning | -11.3 (23.7) | -11.4 (24.0) | -2.2 (17.4)
  Emotional: number analyzed (Participants) | 62 | 66 | 69
  Emotional | 5.4 (17.1) | 3.5 (21.4) | 1.3 (14.0)
  Cognitive: number analyzed (Participants) | 62 | 66 | 69
  Cognitive | 0.5 (12.4) | -2.0 (15.6) | -1.4 (11.0)
  Social Functioning: number analyzed (Participants) | 62 | 66 | 69
  Social Functioning | -8.3 (18.8) | -3.5 (16.7) | -0.7 (12.6)
  Fatigue: number analyzed (Participants) | 62 | 66 | 69
  Fatigue | 13.6 (23.2) | 13.9 (22.6) | 4.0 (12.8)
  Nausea/Vomiting: number analyzed (Participants) | 62 | 66 | 69
  Nausea/Vomiting | 11.8 (17.7) | 9.6 (12.4) | 2.7 (7.4)
  Pain: number analyzed (Participants) | 62 | 66 | 69
  Pain | 4.8 (19.9) | 3.5 (19.3) | 2.9 (16.7)
  Dyspnea: number analyzed (Participants) | 62 | 66 | 69
  Dyspnea | 1.1 (19.1) | 0.5 (19.8) | -1.0 (12.7)
  Insomnia: number analyzed (Participants) | 62 | 66 | 69
  Insomnia | -1.1 (19.1) | 0.5 (29.5) | -1.9 (22.1)
  Appetite Loss: number analyzed (Participants) | 61 | 66 | 69
  Appetite Loss | 16.9 (28.3) | 16.9 (27.5) | 1.9 (15.0)
  Constipation: number analyzed (Participants) | 61 | 65 | 69
  Constipation | 22.4 (31.5) | 16.9 (31.2) | 1.9 (15.0)
  Diarrhea: number analyzed (Participants) | 62 | 66 | 69
  Diarrhea | 18.3 (29.4) | 27.8 (25.9) | 0.0 (15.1)
  Financial Impact: number analyzed (Participants) | 60 | 66 | 69
  Financial Impact | -2.8 (19.7) | 2.0 (18.4) | 0.0 (11.4)

6. Secondary Outcome: Pharmacokinetics (PK): Apparent Clearance of Abemaciclib
Description: Abemaciclib apparent clearance (CL/F) was calculated by population nonlinear mixed effects modeling (NONMEM) using all available data spanning cycles 1 and cycles 3-5.
Time Frame: Cycle(C)1, Day(D)1: 2 to 4 Hours (Hrs) Postdose; C1D14: 4 Hrs Postdose, 7 Hrs Postdose; C3D1: Predose, 3 Hrs Postdose, C4D1 & C5D1, Predose, C5D28: Predose, 3 Hrs Postdose
Population: All randomized participants who received at least one dose of abemaciclib across cycles 1 and cycles 3-5. The results are summarized by the original randomized arms of cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour (L/h)
Groups:
- Abemaciclib: Cycle 1 participants received 150 mg of abemaciclib orally Q12H for 2 weeks.
  All participants received 150 mg of abemaciclib orally Q12H plus 1 mg of anastrozole QD for an additional 14 weeks (post cycle 1).
  Total treatment duration was 16 weeks.
- Anastrozole: Cycle 1 participants received 1 mg of anastrozole orally QD for 2 weeks.
  All participants received 150 mg of abemaciclib orally Q12H plus 1 mg of anastrozole orally QD for an additional 14 weeks (post cycle 1).
  Abemaciclib PK samples were collected during cycles 3-5.
  Total treatment duration was 16 weeks.
  The data presented in this cohort is for abemaciclib PK following cycles 3-5.
Arm/Group | Abemaciclib + Anastrozole | Abemaciclib | Anastrozole
Number analyzed (Participants) | 74 | 75 | 74
Liters/hour (L/h) | 24.0 (32) | 19.1 (55) | 24.4 (61)

7. Secondary Outcome: PK: Apparent Volume of Distribution of Abemaciclib
Description: Abemaciclib apparent volume of distribution was calculated by population NONMEM using all available data spanning cycles 1 and cycles 3-5.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | Abemaciclib + Anastrozole | Abemaciclib | Anastrozole
Number analyzed (Participants) | 74 | 75 | 74
Liters (L) | 941 (53) | 720 (58) | 758 (49)

ADVERSE EVENTS:
Time Frame: Up to 24 Weeks
Description: All randomized participants who received at least one dose of study drug.
Groups:
- Abemaciclib + Anastrozole Cycle 1: Participants were given 150 mg of abemaciclib orally Q12H plus 1 mg of anastrozole orally QD for 2 weeks.
  All participants received 150 mg of abemaciclib orally Q12H plus 1 mg of anastrozole orally QD for an additional 14 weeks.
  Total treatment duration was 16 weeks.
- Abemaciclib Cycle 1: Participants received 150 mg of abemaciclib orally QD for 2 weeks.
  All participants received 150 mg of abemaciclib orally Q12H plus 1 mg of anastrozole orally QD for an additional 14 weeks.
  Total treatment duration was 16 weeks.
- Anastrozole Cycle 1: Participants received 1 mg of anastrozole orally Q12H for 2 weeks.
  All participants received 150 mg of abemaciclib orally Q12H plus 1 mg of anastrozole QD for an additional 14 weeks.
  Total treatment duration was 16 weeks.
  .
- Abemaciclib + Anastrozole Cycle 2 and Beyond: Combination Therapy: All participants received 150 mg of abemaciclib orally Q12H plus 1 mg of anastrozole orally QD for an additional 14 weeks.
  Total treatment duration was 16 weeks.
Arm/Group | Abemaciclib + Anastrozole Cycle 1 | Abemaciclib Cycle 1 | Anastrozole Cycle 1 | Abemaciclib + Anastrozole Cycle 2 and Beyond
Serious Adverse Events (participants affected / at risk) | 1/74 | 1/75 | 0/74 | 16/217
Other Adverse Events (participants affected / at risk) | 62/74 | 58/75 | 17/74 | 189/217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib + Anastrozole Cycle 1 (N=74) | Abemaciclib Cycle 1 (N=75) | Anastrozole Cycle 1 (N=74) | Abemaciclib + Anastrozole Cycle 2 and Beyond (N=217)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib + Anastrozole Cycle 1 (N=74) | Abemaciclib Cycle 1 (N=75) | Anastrozole Cycle 1 (N=74) | Abemaciclib + Anastrozole Cycle 2 and Beyond (N=217)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 27 (31)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 0 (0) | 19 (22)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 45 (58)
Abdominal pain (Gastrointestinal disorders) | 13 (15) | 7 (7) | 2 (2) | 30 (34)
Constipation (Gastrointestinal disorders) | 27 (27) | 26 (30) | 5 (5) | 50 (62)
Diarrhoea (Gastrointestinal disorders) | 31 (34) | 29 (33) | 2 (2) | 101 (162)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 5 (5) | 0 (0) | 7 (8)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 1 (1) | 0 (0) | 7 (7)
Nausea (Gastrointestinal disorders) | 19 (19) | 15 (15) | 2 (2) | 67 (75)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 19 (21)
Vomiting (Gastrointestinal disorders) | 5 (6) | 1 (1) | 0 (0) | 25 (32)
Fatigue (General disorders) | 19 (20) | 17 (18) | 3 (4) | 62 (70)
Alanine aminotransferase increased (Investigations) | 4 (4) | 1 (1) | 0 (0) | 26 (27)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 1 (1) | 0 (0) | 22 (23)
Blood creatinine increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 14 (15)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 15 (17)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 13 (13) | 0 (0) | 33 (36)
Dizziness (Nervous system disorders) | 1 (1) | 5 (5) | 1 (1) | 8 (10)
Dysgeusia (Nervous system disorders) | 4 (4) | 5 (5) | 0 (0) | 17 (18)
Headache (Nervous system disorders) | 3 (3) | 5 (5) | 0 (0) | 16 (17)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 12 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 20 (21)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 22 (24)
Hot flush (Vascular disorders) | 3 (3) | 2 (2) | 5 (5) | 19 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less